CLINICAL TRIAL: NCT03269318
Title: Feasibility of a Personalised Medicine Clinic for Children With Asthma Aged 5-11 Years
Brief Title: PRISTINE - Personalised Approach to Improve aSThma prescrIbing iN childrEn
Acronym: PRISTINE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change to Primary Endpoint resulted in development of new protocol
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 183898
Record Dates: First submitted 2017-07-11; First posted 2017-08-31 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Salmeterol Xinafoate; Theophylline; Steroids

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to one of two groups as per block randomisation, with no stratification or minimisation to Group 1; Personalised Medicine who will be prescribed controller medication based on genetic test, Arg/Arg or Arg/Gly - montelukast (LTRA) or Gly/Gly -salmeterol (LABA). While Group 2, Standard Care will be prescribed controller medication based on guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised Medicine (Experimental): Personalised Medicine who will be prescribed controller medication based on genetic test, Arg/Arg or Arg/Gly - montelukast (LTRA) or Gly/Gly -salmeterol (LABA).
  Interventions: Drug: Montelukast or Salmeterol or Theophylline or Steroid
- Standard Care (No Intervention): Standard of care (Standard Care will be prescribed controller medication based on guidelines)

INTERVENTIONS:
Drug: Montelukast or Salmeterol or Theophylline or Steroid — Medication will be patient specific according to their current medication, clinical symptoms and genotype. It will be from a choice of; leukotriene receptor antagonist (montelukast), long-acting beta2 agonist (salmeterol), theophylline or increase dose of inhaled steroid.
  Arms: Personalised Medicine

SUMMARY:
Asthma is one of the most common chronic diseases affecting children in the UK. Poorly controlled asthma manifests with chronic cough, wheeze and shortness of breath which in-turn has a significant negative impact on a child's quality of life, interfering with sleep, impairing exercise ability and resulting in frequent school absences and hospital admissions.

Management of paediatric asthma in the UK is directed by the British Thoracic Society (BTS) Guidelines, which recommend a stepwise (one to five) treatment plan. Step three of the management guideline for children aged 5-12 years of age recommends the addition of the preventer inhaled medication, including long-acting β2 agonists such as salmeterol. However, there is a wide variation in response to this medication with approximately one in seven people, with a specific genetic change, found to have an increase in asthma symptoms in association with the use of thisiss medication. A related medicine, formoterol, is used less commonly in children with asthma.

In this study, the investigators will aim to identify children with asthma whose symptoms are poorly controlled on inhaled long-acting beta2 agonists. Via a simple saliva test, the investigators will identify the presence or absence of the specific genetic change potentally influencing the effectiveness of treatment with salmeterol or related longacting beta2 agonists thus enabling the investigators to recommend either salmeterol or an alternative medication for the treatment plan such as montelukast. The investigators will randomise the patients into two groups; to receive "personalised care" where the choice of controller medication would be based on the child's gene test results and predicted response to long-acting beta2 agonists, or "standard care" following the BTS guidelines at the clinician's discretion without knowledge of the gene test results. The investigators aim to measure whether this individualized approach to asthma prescribing results in improved control of asthma symptoms and overall quality of life. Targeting treatment to a child's specific genetic make-up is a concept known as "personalised medicine".

DETAILED DESCRIPTION:
Asthma is a common chronic illness in children and young people. It affects, for example, an average of two children in every UK classroom. Initial treatment usually consists of salbutamol used on demand at step 1 of British Thoracic Society (BTS) guidelines. At step 2, regular anti-inflammatory 'controller' therapy starts with the regular use of inhaled corticosteroids such as beclomethasone. Therapeutic efficacy with inhaled steroids usually peaks around 400 micrograms per day of beclomethasone (or equivalent). With inadequate asthma control at step 2, inhaled long-acting β2 agonists (LABA) such as salmeterol, or leukotriene receptor antagonists (LTRA) such as montelukast are added or inhaled corticosteroids are increased; this represents BTS step 3 for asthma management.

Overall, in children with asthma managed on step 3, salmeterol appears to provide better asthma control than montelukast in the setting of a randomized controlled trial. However, in real life, the efficacy of salmeterol at step 3 for improving asthma control in individual children appears rather variable, and some children continue to experience day-to-day symptoms and exacerbations.

In this study of 1182 UK children and young adults (4-22 years), 50% of those on regular salmeterol experienced asthma exacerbations over a 6-month period, and 18% required inhaled salbutamol at least daily for symptom relief. Indeed, the investigators reported a step-wise increase in the risk of asthma attacks related to each copy of the Arg16 allele on the β2 receptor gene (1.7-fold) in asthmatic children and young adults exposed to regular salmeterol in conjunction with inhaled corticosteroids. This led the investigators to hypothesize that, contrary to the observations on the overall population of children and young adults where salmeterol is superior in efficacy to montelukast at step 3, those possessing susceptible Arg16 β2 receptor genotype may experience better asthma control with the addition of montelukast rather than salmeterol as second-line controller medication, in addition to inhaled corticosteroids. As such the investigators elected to identify from the database those children with two copies of the Arg16 polymorphism [i.e. homozygous Arg genotype (∼15% of overall population) who would potentially be at greatest risk]. The mechanism for worse control with regular salmeterol involves a greater susceptibility to agonist-induced down-regulation and uncoupling of airway β2 receptors and associated sub-sensitivity of response in the Arg16 genotype.

The investigators therefore performed a proof-of-concept randomized controlled trial to determine whether genetically susceptible children with homozygous Arg16 genotype experience superior long-term asthma control with montelukast compared with salmeterol when used as tailored second-line controller therapy as add-on to the inhaled steroid fluticasone. The purpose of this preliminary study was to provide evidence to support the potential for personalised medicine based on the individual genotype to improve asthma-related quality-of-life and control. This study was published in 2013, and represents the first prospective randomized controlled study in children with asthma that addresses personalised medicine based on genotype. The results of this study showed that in children expressing the homozygous Arg 16 genotype, in comparison with salmeterol, adding montelukast to inhaled fluticasone significantly improved asthma-related quality-of-life and clinical symptoms, while reducing school absences and inhaled reliever use. The relative benefits of montelukast in comparison with salmeterol became evident within the first 3 months and persisted throughout the whole year.

Subsequently, the investigators used Pubmed to search the Medline database for other randomised controlled trials comparing the effects of salmeterol (or other long-acting beta2 agonist) with montelukast (or other leukotriene antagonist) within the context of Arg/Gly variation, in children with asthma. No studies could be identified. In particular, there are no trials in either adults or children that have studied quality-of-life, which is a key outcome of interest in the context of asthma-related disability, and which is often unrelated to outcomes such as lung function. This led to the development of the Personalised Medicine for Asthma Control (PACT)-study, a randomised controlled trial to determine if personalised medicine improves quality of life and asthma control in 12-18 years olds. Results of this trial when published, will provide more conclusive evidence as to the effectiveness of personalised medicine in this age group. However, there is an absence of trials in a younger age group of children with asthma (5-11 years) and no evidence to determine if a personalised medicine clinic is feasible within a hospital setting, which underscores the need for this study.

There is an absence of trials in a younger age group of children with asthma (5-11 years) and no evidence to determine if a personalised medicine clinic is feasible within a hospital setting and this underscores the need for this study.

This research proposes two stages of work and has two main objectives:

1. Feasibility study: Conduct a feasibility study to determine important parameters (standard deviation of outcomes, recruitment and retention) to inform the design of a definitive randomised controlled trial

   Research questions:
   1. Are children with asthma and their parents willing to be recruited and randomised to a trial of genotyping and personalised management for asthma?
   2. Are there retention issues? If yes, at what stages did these occur? What were the reasons?
   3. Are follow-up data complete?
   4. Can the intervention (genotyping plus medication) be delivered with sufficient fidelity?
   5. Is there sufficient evidence for scaling up to a definitive randomised controlled trial?
   6. What sample size is needed to power a full scale randomised controlled trial?
   7. Are there any safety issues or adverse events?
   8. What are the associated costs of running a personalised asthma clinic and is it cost effective?
2. Qualitative aspect: Assess the acceptability of a personalised asthma clinic for children with asthma

Research questions:

1. How acceptable do children with asthma and their parents find genotyping and the personalised approach? How does this compare with their views on acceptability of conventional clinics?
2. Was there any aspect of genotyping and personalised medicine clinic which children with asthma and their parents thought was particularly good or worked well?
3. Was there any aspect of genotyping and personalised medicine clinic which children with asthma and their parents thought was particularly bad or difficult?
4. How satisfied were children with asthma and their parents with the genotyping and personalised medicine clinic?
5. How did the genotyping and personalised medicine clinic differ from usual care?
6. What would encourage other children with asthma and their parents to participate in a genotyping and personalised medicine clinic?
7. What would participants change about the personalised clinic?
8. How has the genotyping and personalised medicine clinic impacted on the child and their parent?
9. Were there any outcomes which weren't measured which should have been?
10. What did the health professionals involved think about the clinic? (in primary and secondary care)

Two arm, randomised controlled feasibility trial of genotyping and personalised medicine versus usual care with qualitative aspect to assess acceptability and impact.

The genotyping and personalised medicine clinic is based in the Royal Alexandra Children's Hospital in Brighton, England. Participants are referred to the research team by their health care professional (primary and secondary care).

The intervention and follow up period will last 4 months per participant. Outcomes will be measured at baseline and 3-months.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Guardian/Participant is willing and able to give informed consent/assent
* Physician-diagnosed asthma that is inadequately controlled as per view of doctor (for example, history of at least two emergency visits to GP or hospital over the previous year, frequent use of blue inhaler (three times or more per week))
* Aged 5-11 years (inclusive)
* Children who are already on at least 400 micrograms per day inhaled beclomethasone or equivalent and hence ready to be prescribed inhaled long-acting beta2 agonists and/or other add-on medication or are already on inhaled long-acting beta2 agonists and/or other add-on medication

Exclusion Criteria:

* Parent/Guardian/Participant is unwilling or unable to give informed consent/assent
* Known contraindication to montelukast or salmeterol
* Other known significant airway or lung disease (e.g. chronic lung disease of prematurity, cystic fibrosis or congenital airway abnormalities) or other co-existing serious disease such as congenital cardiac disease
* Poor inhaler technique and/or history of poor adherence on checking following standard procedure at the clinic
* Participating in another clinical trial (other than observational trials and registries) concurrently or within 30 days prior to screening for entry into this study

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Are children with asthma and their parents willing to be recruited and randomised to a trial of genotyping and personalised management for asthma? Qualitative interview | Baseline to 3 months
  Recruitment rates will be measured as rate of invited participants who are eligible and consenting and will be reported in a Consolidated Standards of Reporting Trials (CONSORT) participant flowchart.
Are there retention issues? If yes, at what stages did these occur? What were the reasons? Qualitative interview | Baseline to 3 months
  Acceptability of allocation procedures will be assessed by examining reasons for dropout in discontinuing participants and comparing attrition rates between the two study groups and between participants who did and did not receive their preferred allocation. Attrition rates will be established as discontinuation of intervention and loss to follow-up measurement for both groups
Are follow-up data complete? | Baseline to 3 months
  Suitability of outcome measures will be evaluated based on completion rates and rates of missing data
Acceptability of personalised approach | Baseline to 3 months
  All participants and their parents/guardians will be invited to have a semi-structured interview with a member of the research team in order to discuss their experiences of living with and managing their asthma. To enhance communication and ensure the child's perspective is captured, children will be invited to make a drawing of what it is like to have asthma and what it feels like when they take their asthma medication. The research team interviewing will then discuss the drawings (as a visual cue) in simple language with each child to understand what the child means.

SECONDARY OUTCOMES:
Childhood Asthma Control Test | Baseline to 3 months
  The Childhood Asthma Control Test (C-ACT) [10], a 7-item validated questionnaire capturing the frequency of asthma symptoms and their effect on daily function in children 4 to 11 years of age. It uses a 4-point Likert scale with higher scores indicating better control. The C-ACTuses a single cut point of a score of ≤19 to identify children whose asthma is not well controlled.
Lung Function | Baseline to 3 months
  Lung function will be measured by a nurse trained in collecting spirometry data in the Royal Alexandra Children's Hospital. Measure of PEF (litres/second), FEV1 (litres) and FVC (litres)
Days unable to complete usual activities | Baseline to 3 months
  Participants and parents will be asked to report how many days in the last month they have been unable to complete usual activities as a result of their asthma.
Use of medication | Baseline to 3 months
  Number of courses of oral corticosteroids for asthma and any other medication use will be recorded.
Use of health services | Baseline to 3 months
  Participants and parents will be asked to report how many times they have had to see their GP or asthma nurse (outside of routine asthma review), been to A&E or been admitted to hospital as a result of their asthma.
Beliefs about medicine questionnaire | Baseline to 3 months
  The Beliefs About Medicine Questionnaire (BMQ) [11] is an 18-item validated questionnaire which will capture parental beliefs about asthma, asthma medication and how these may have affected their child's life. Respondents indicate their degree of agreement with each individual statement about medicines on a 5-point Likert scale, (1=strongly disagree to 5=strongly agree). Scores obtained are summed to give a scale score with higher scores indicating stronger beliefs.
Experience of service | 3 month visit
  At the final follow up, participants and parents will be asked to comment on their experience of the service received in the personalised medicine clinic. The validated Commission for Health Improvement Experience of Service Questionnaire will be used as the outcome measure [12]. The ESQ consists of 12 items rated on a 3-point Likert scale (3=Certainly True to 1=Not true) and three free-text sections looking at what the respondent liked about the clinic, what they felt needed improving, and any other comments. Higher scores indicate more positive experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Prof Mukhopadhyay, Principal Investigator — Brighton and Sussex University Hospital NHS Trust
Locations (1):
- BrightonNHS, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided